CLINICAL TRIAL: NCT05093829
Title: A Phase 3 Trial to Evaluate the Safety, Immunogenicity, and Non-Interference With Concomitant Routine Vaccines, of a Meningococcal Serogroup ACYWX Conjugate Vaccine (NmCV-5) in Comparison With MenACWY-TT Conjugate Vaccine in Healthy Malian Infants
Brief Title: Meningococcal Serogroup ACYWX Conjugate Vaccine in Comparison With MenACWY-TT Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Wilbur Chen, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EUCC-DMID-20-0024; UM1AI148689 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Meningitis
Keywords: vaccine; meningococcal; Neisseria meningitidis; conjugate meningococcal vaccine; meningococcal serogroup X
MeSH Terms: conditions — Meningitis | interventions — NmCV-5 vaccine; tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vaccination at 9 months of age with NmCV-5 (Experimental): Infant participants randomized to receive the NmCV-5 meningococcal vaccination at 9 months of age, while receiving the current Mali EPI schedule of vaccines.
  Interventions: Biological: NmCV-5
- Vaccination at 9 months of age with MenACWY-TT (Active Comparator): Infant participants randomized to receive the MenACWY-TT meningococcal vaccination at 9 months of age, while receiving the current Mali EPI schedule of vaccines.
  Interventions: Biological: MenACWY-TT
- Vaccination at 15 months of age with NmCV-5 (Experimental): Infant participants randomized to receive the NmCV-5 meningococcal vaccination at 15 months of age, while receiving the current Mali EPI schedule of vaccines.
  Interventions: Biological: NmCV-5
- Vaccination at 15 months of age with MenACWY-TT (Active Comparator): Infant participants randomized to receive the MenACWY-TT meningococcal vaccination at 15 months of age, while receiving the current Mali EPI schedule of vaccines.
  Interventions: Biological: MenACWY-TT

INTERVENTIONS:
Biological: NmCV-5 — NmCV-5 is a pentavalent meningococcal (A, C, Y, W, X) polysaccharideconjugate vaccine composed of capsularpolysaccharides (PS) from Neisseria meningitidis serogroups A, C, Y, W, and X individually conjugated to a protein carrier, either mutant diphtheria toxoid (CRM197) or tetanus toxoid (TT).
  Arms: Vaccination at 15 months of age with NmCV-5; Vaccination at 9 months of age with NmCV-5
Biological: MenACWY-TT — MenACWY-TT (the comparator meningococcal vaccine) is a WHO-PQ quadrivalent meningococcal (A, C, Y, W) polysaccharide-conjugate vaccine manufactured by Pfizer.
  Other Names: Nimenrix
  Arms: Vaccination at 15 months of age with MenACWY-TT; Vaccination at 9 months of age with MenACWY-TT

SUMMARY:
Infants aged 9 months will be randomized to receive a meningococcal vaccine at 9 months or 15 months. Infants randomized to the 9-month age group will be further randomized in a 2:1 ratio to receive a single dose of the experimental meningococcal vaccine (NmCV-5) or a single dose of the comparator meningococcal vaccine (MenACWY-TT). Prospectively identified and consented infants randomized to the 15-month age group will return when aged 15 months and will be randomized in a 2:1 ratio to receive a single dose of NmCV-5 or a single dose of MenACWY-TT.

DETAILED DESCRIPTION:
Meningococcal meningitis, caused by invasive strains of Neisseria meningitidis, is a major public health concern because of its considerable morbidity and mortality in sub-Saharan Africa. Case fatality during meningococcal meningitis epidemics can surpass 15%, and rates of permanent sequelae among meningitis survivors in Africa are twice as high as they are in high income countries. Because of the fulminant clinical course of invasive bacterial meningitis and difficulties in access to care in the African meningitis belt, prevention by vaccination is the optimal way to reduce meningococcal meningitis morbidity and mortality. Before 2010, serogroup A meningococcal strains were routinely responsible for the majority (70-96%) of invasive meningococcal disease in sub-Saharan Africa. And annual epidemic could be associated with an incidence of meningococcal disease which could range between 100-1000 cases per 100,000 persons in any given year.

Progressive introduction of MenAfriVac since 2010 has resulted in a substantial reduction in cases of serogroup A meningococcal disease. However, regular large-scale epidemics due to serogroups C, W and X remain common in the African meningitis belt. An affordable and scalable pentavalent meningococcal conjugate vaccine (NmCV-5) has been developed by Serum Institute of India Pvt. Ltd. (SIIPL), the manufacturer of MenAfriVac. NmCV-5 is designed to protect against serogroups A, C, W, Y and X. The immediate goal for the clinical development of NmCV-5 is for WHO Pre-Qualification (WHO-PQ), to enable the vaccine to be used in the Meningitis Belt of sub-Saharan Africa.

This trial will evaluate a single dose of NmCV-5 administered at either 9 months or 15 months of age, time points in the Expanded Program on Immunization (EPI) schedule when meningococcal vaccine is most likely to be administered. Infants aged 9 months will be randomized to receive a meningococcal vaccine at 9 months or 15 months. Infants aged 9 months (eligibility 9-11 months) and randomized to the 9-month age group will be randomized in a 2:1 ratio to receive a single dose of NmCV-5 or a single dose of MenACWY-TT. Prospectively identified and consented infants randomized to the 15-month age group will return when aged 15 months (eligibility 15-17 months) and will be randomized in a 2:1 ratio to receive a single dose of NmCV-5 or a single dose of MenACWY-TT. "Enhanced" EPI vaccines will be co-administered and will consist of 2-doses of a measles-containing vaccine administered at 9 months and 15 months and a single dose of yellow fever vaccine administered at 9 months.

This study protocol is designed to provide evidence that concomitant vaccination with NmCV-5 will not significantly affect the immune responses of infants to their normally scheduled EPI vaccines. This study has been specifically designed to provide information at two distinct timepoints, 9 months and 15 months. The current Mali EPI schedule consists of a measles only vaccine, yellow fever vaccine, and MenA vaccine at 9 months of age; there is no 15 months of age EPI vaccine visit and typically only a single dose of a measles-containing vaccine is administered. However, to satisfy the conditions for WHO-PQ, study participants will receive two doses of a measles-containing vaccine, at 9-months and 15-months. Furthermore, the noninferiority evaluation must include an assessment of the rubella vaccine responses. These modifications to the standard Malian EPI schedule provide a level-of-care that is higher than the current standard-of-care for the general population. Within the context of this study, the researchers will refer to this as an "enhanced" EPI schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children between 9 months and 11 months old inclusive.
2. Parent(s)/legal guardian(s) have provided written informed consent, after the nature of the study has been explained according to local regulatory requirements.
3. The investigator believes that their parent(s)/guardian(s) will be available for all the subjects visits and will comply with the requirements of the protocol (e.g., timely reporting of adverse events).
4. Individual is in good health as determined by medical history, physical examination, and clinical judgement of the investigator.
5. Individual has completed their local infant EPI vaccines, not including 9-month EPI vaccines (at the 9-month visit) or 15- month EPI vaccines (at the 15-month visit). A birth dose of oral polio vaccine is not required.

Exclusion Criteria:

1. History of receipt of any meningococcal vaccine.
2. Has received a measles-containing vaccine.
3. Current or previous, confirm or suspected disease caused by N. meningitidis.
4. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrolment or study vaccination (for the 15-month age group).
5. History of severe allergic reactions after previous vaccinations or hypersensitivity to any study vaccine component including tetanus, diphtheria and mutant diphtheria toxoid (CRM197).
6. Acute or chronic, clinically significant pulmonary, cardiovascular, metabolic, neurological, hepatic, or renal functional abnormality, as determined by medical history or physical examination.
7. Any confirmed or suspected condition with impaired or altered function of the immune system (e.g., immunodeficiency, autoimmune conditions, malnutrition).
8. Have any bleeding disorder which is considered a contraindication to intramuscular injection or blood draw.
9. Severe acute malnutrition. Note: a weight-for-length Z-score of less than -3 satisfies this exclusion criteria.
10. History of either hepatitis B or hepatitis C virus infection, human immunodeficiency virus infection, or hereditary immunodeficiency.
11. Presence of major and clinically significant congenital defects.
12. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within three months prior to the study vaccination or planned use throughout the study period (for corticosteroids, this means prednisone, or equivalent, ≥ 0.5 mg/kg per day. Inhaled, intranasal, and topical steroids are allowed).
13. Administration of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 3 months or planned use throughout the study period.
14. Administration of any vaccine within 14 days prior to enrolment in the study or planned administration of any vaccine within 14 days before or after study vaccination.
15. Use of any investigational or non-registered drug or vaccine within 28 days prior to the administration of study vaccine or planned during the study.
16. Malaria infection as confirmed by a Rapid Diagnostic Test. Note: subjects positive at screening may be treated for malaria as per national guidelines outside of the study, and if the subject remains eligible, vaccinated no earlier than 5 days after completing treatment.
17. Individuals who are close family member* of individuals conducting this study. *defined as a child with direct genetic relationship to a member of the study team.
18. Have experienced a moderate or severe acute infection and/or fever (defined as temperature ≥ 37.5°C) within 3 days prior to enrolment or study vaccination.
19. Have received systemic antibiotic treatment within 3 days prior to enrolment or study vaccination.
20. Non-residence in the study area or intent to move out within six months.
21. Any condition which, in the opinion of the investigator, might post additional risk to the subject due to participation in the study.

Ages: 9 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1325 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2025-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilbur Chen, MD, MS, Study Chair — University of Maryland, Baltimore; Karen Kotloff, MD, Study Director — University of Maryland, Baltimore
Locations (1):
- Centre pour le Developpement des Vaccins du Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diallo F, Haidara FC, Tapia MD, Dominguez Islas CP, Alderson MR, Hausdorff WP, Martellet L, Hosken N, Kapse D, Kulkarni PS, Townsend-Payne K, Vanni F, Posavad CM, Sow SO, Kotloff KL, Chen WH; NmCV-5 EPI study team. Safety and immunogenicity of a pentavalent meningococcal conjugate vaccine targeting serogroups A, C, W, Y, and X when co-administered with routine childhood vaccines at ages 9 months and 15 months in Mali: a single-centre, double-blind, randomised, controlled, phase 3, non-inferiority trial. Lancet. 2025 Mar 29;405(10484):1069-1080. doi: 10.1016/S0140-6736(25)00046-7. Epub 2025 Mar 11. PMID 40086461
- [Derived] Stephens DS. Global Control of Meningococcal Disease. N Engl J Med. 2023 May 25;388(21):2003-2005. doi: 10.1056/NEJMe2301698. No abstract available. PMID 37224203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Mali, enrollment began March 24, 2022, and all follow up at Day 29 was complete by March 10, 2023.
Pre-assignment Details: 1331 participants were assessed for eligibility and 6 were ineligible and excluded. 1325 participants received step 1 randomization to Group 1 (meningococcal vaccination at 9 months of age, n=602) or Group 2 (meningococcal vaccination at 15 months of age, n=723). 1202 participants received step 2 randomization to meningococcal vaccine study arm, and 123 Group 2 participants were excluded due to lost to follow-up or ineligibility or Group 2 target (n=600) met.
Groups:
- Vaccination at 9 Months of Age With NmCV-5: Infant participants randomized to receive the NmCV-5 meningococcal vaccination at 9 months of age, while receiving concomitant EPI vaccines.
  NmCV-5: NmCV-5 is a pentavalent meningococcal (A, C, Y, W, X) polysaccharideconjugate vaccine composed of capsularpolysaccharides (PS) from Neisseria meningitidis serogroups A, C, Y, W, and X individually conjugated to a protein carrier, either mutant diphtheria toxoid (CRM197) or tetanus toxoid (TT).
- Vaccination at 9 Months of Age With MenACWY-TT: Infant participants randomized to receive the MenACWY-TT meningococcal vaccination at 9 months of age, while receiving concomitant EPI vaccines.
  MenACWY-TT: MenACWY-TT (the comparator meningococcal vaccine) is a WHO-PQ quadrivalent meningococcal (A, C, Y, W) polysaccharide-conjugate vaccine manufactured by Pfizer.
- Not Vaccinated But Randomized to Vaccination at 15 Months of Age: Infant participants receiving step 1 randomization to Group 2 (meningococcal vaccination at 15 months of age) and discontinued from the study prior to step 2 randomization and meningococcal vaccination because Group 2 vaccination target was met.
- Vaccination at 15 Months of Age With NmCV-5: Infant participants randomized to receive the NmCV-5 meningococcal vaccination at 15 months of age, while receiving concomitant EPI vaccines.
  NmCV-5: NmCV-5 is a pentavalent meningococcal (A, C, Y, W, X) polysaccharideconjugate vaccine composed of capsularpolysaccharides (PS) from Neisseria meningitidis serogroups A, C, Y, W, and X individually conjugated to a protein carrier, either mutant diphtheria toxoid (CRM197) or tetanus toxoid (TT).
- Vaccination at 15 Months of Age With MenACWY-TT: Infant participants randomized to receive the MenACWY-TT meningococcal vaccination at 15 months of age, while receiving concomitant EPI vaccines.
  MenACWY-TT: MenACWY-TT (the comparator meningococcal vaccine) is a WHO-PQ quadrivalent meningococcal (A, C, Y, W) polysaccharide-conjugate vaccine manufactured by Pfizer.
Period: Step 1 Randomization
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Not Vaccinated But Randomized to Vaccination at 15 Months of Age | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Started | 401 | 201 | 123 | 400 | 200
Completed | 401 | 201 | 123 | 400 | 200
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Step 2 Randomization
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Not Vaccinated But Randomized to Vaccination at 15 Months of Age | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Started | 401 | 201 | 123 | 400 | 200
Completed | 401 | 201 | 0 | 400 | 200
Not Completed | 0 | 0 | 123 | 0 | 0
Not completed — Lost to follow-up, ineligibility, or Group 2 target met | 0 | 0 | 123 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two participants refused the meningococcal vaccination (1 participant in each vaccine study arm in Group 1, meningococcal vaccination at 9 months of age) and were excluded from the mITT analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT | Total
Number analyzed (Participants) | 400 | 200 | 400 | 200 | 1200
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.3 (0.5) | 9.3 (0.5) | 9.3 (0.5) | 9.2 (0.5) | 9.3 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 101 | 201 | 108 | 613
  Male | 197 | 99 | 199 | 92 | 587
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 400 | 200 | 400 | 200 | 1200
Region of Enrollment [Number; unit: participants]
  Mali | 400 | 200 | 400 | 200 | 1200
Participant Height/Length [Mean (Standard Deviation); unit: cm] | 70.1 (2.4) | 70.2 (2.9) | 70.0 (2.6) | 69.9 (2.5) | 70.0 (2.6)
Participant weight [Mean (Standard Deviation); unit: kg] | 8.1 (1.0) | 8.0 (1.1) | 8.1 (1.0) | 8.0 (0.9) | 8.0 (1.0)
Participant Length-for-weight z-score [Mean (Standard Deviation); unit: z-score] — This is a WHO standardized method to classify a child's nutritional status where a Z-score of 0 (zero) represents the global population mean score of the weight divided by height for age. A Z-score of "+1" or "-1" is a value that is one standard deviation above or below the mean where Z-scores below the mean demonstrate a lower/poorer developmental/nutritional status than the rest of the world. The use of anthropometry based on this Z-score is commonly used to classify malnutrition, as follows -1 to -1.9: mild malnutrition, -2.0 to -2.9: moderate malnutrition and ≥ -3: severe malnutrition.
  z-score | -0.4 (1.1) | -0.5 (1.1) | -0.4 (1.1) | -0.5 (1.0) | -0.4 (1.1)
Participant Body Temperature [Mean (Standard Deviation); unit: Celcius] | 36.0 (0.4) | 36.0 (0.4) | 36.1 (0.4) | 36.1 (0.4) | 36.0 (0.4)
Participant Heart Rate, Pulse [Mean (Standard Deviation); unit: beats/minute] | 112.6 (4.0) | 112.8 (4.3) | 111.8 (3.7) | 112.2 (3.9) | 112.3 (3.9)
Participant Rate of Respiration [Mean (Standard Deviation); unit: breaths/minute] | 25.4 (2.9) | 25.6 (2.7) | 25.4 (2.8) | 25.2 (2.8) | 25.4 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroprotection for Meningitis Serogroups A, C, W and Y
Description: Null hypothesis: The immune response to meningitis serogroup "S" at Day 29 elicited by one dose of NmCV-5 is inferior to the immune response elicited by one dose of MenACWY-TT.
  Alternative hypothesis: The immune response to meningitis serogroup "S" at Day 29 elicited by one dose of NmCV-5 is non-inferior, by a pre-specified margin, to the immune response elicited by one dose of MenACWY-TT, where "S" denotes one of the meningitis serogroups: A, C, W or Y. Endpoints are the seroprotective response at Day 29 to serogroups A, C, W and Y in the NmCV-5 arm and seroprotective response at Day 29 to serogroups A, C, W and Y in the MenACWY-TT arm with seroprotective response defined as serogroup specific rSBA antibody titers ≥ 8.
  Non-inferiority comparisons are made between study vaccination arms within each study age group (9 months or 15 months of age).
  Proportions and difference in proportions are reported as percentages (number of infants per 100).
Time Frame: Measured from time of meningococcal vaccination to blood sample collection at Day 29 visit. Follow-up time to Day 29 visit blood specimen collection was a mean (s.d.) of 30.9 (2.8) days.
Population: All participants included in the Per Protocol (PP) Analysis Set which includes eligible participants receiving step 1 and 2 randomizations, the randomized meningococcal vaccination in the appropriate age group window with the scheduled EPI vaccinations, and who had a blood specimen collected in the appropriate window around the Day 29 visit and a successful rSBA value provided by the laboratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 373 | 191 | 367 | 182
Participants
  Participants with seroprotective response against meningococcal serogroup A: Yes | 373 | 191 | 366 | 180
  Participants with seroprotective response against meningococcal serogroup A: No | 0 | 0 | 1 | 2
  Participants with seroprotective response against meningococcal serogroup C: Yes | 369 | 190 | 358 | 179
  Participants with seroprotective response against meningococcal serogroup C: No | 4 | 1 | 9 | 3
  Participants with seroprotective response against meningococcal serogroup W: Yes | 352 | 186 | 362 | 179
  Participants with seroprotective response against meningococcal serogroup W: No | 21 | 5 | 5 | 3
  Participants with seroprotective response against meningococcal serogroup Y: Yes | 360 | 190 | 364 | 178
  Participants with seroprotective response against meningococcal serogroup Y: No | 13 | 1 | 3 | 4
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup A, the proportion of infants with a seroprotective response to MenACWY-TT is subtracted from the proportion of infants with a seroprotective response to NmCV-5 to determine the difference in proportions; Test type: Non-Inferiority — NmCV-5 will be deemed non-inferior to MenACWY-TT for serogroup A if the lower limit of the 95% confidence interval for the difference in proportion (NmCV-5 minus MenACWY-TT) excludes -0.10 (-10%). Confidence Intervals are calculated using the Miettinen-Nurminen method. Difference in proportions and confidence intervals are reported as percentages (number of infants per 100); Difference in proportions = 0.0, 95% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 2: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in proportions = 0.8, 95% CI 2-sided [-0.6 to 3.7]
Statistical Analysis 3: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup C, the proportion of infants with a seroprotective response to MenACWY-TT is subtracted from the proportion of infants with a seroprotective response to NmCV-5 to determine the difference in proportions; Test type: Non-Inferiority — NmCV-5 will be deemed non-inferior to MenACWY-TT for serogroup C if the lower limit of the 95% confidence interval for the difference in proportion (NmCV-5 minus MenACWY-TT) excludes -0.10 (-10%). Confidence Intervals are calculated using the Miettinen-Nurminen method. Difference in proportions and confidence intervals are reported as percentages (number of infants per 100); Difference in proportions = -0.5, 95% CI 2-sided [-2.3 to 1.9]
Statistical Analysis 4: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 3]; Difference in proportions = -0.8, 95% CI 2-sided [-3.3 to 2.5]
Statistical Analysis 5: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup W, the proportion of infants with a seroprotective response to MenACWY-TT is subtracted from the proportion of infants with a seroprotective response to NmCV-5 to determine the difference in proportions; Test type: Non-Inferiority — NmCV-5 will be deemed non-inferior to MenACWY-TT for serogroup W if the lower limit of the 95% confidence interval for the difference in proportion (NmCV-5 minus MenACWY-TT) excludes -0.10 (-10%). Confidence Intervals are calculated using the Miettinen-Nurminen method. Difference in proportions and confidence intervals are reported as percentages (number of infants per 100); Difference in proportions = -3.0, 95% CI 2-sided [-6.3 to 0.8]
Statistical Analysis 6: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 5]; Difference in proportions = 0.3, 95% CI 2-sided [-1.8 to 3.5]
Statistical Analysis 7: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup Y, the proportion of infants with a seroprotective response to MenACWY-TT is subtracted from the proportion of infants with a seroprotective response to NmCV-5 to determine the difference in proportions; Test type: Non-Inferiority — NmCV-5 will be deemed non-inferior to MenACWY-TT for serogroup Y if the lower limit of the 95% confidence interval for the difference in proportion (NmCV-5 minus MenACWY-TT) excludes -0.10 (-10%). Confidence Intervals are calculated using the Miettinen-Nurminen method. Difference in proportions and confidence intervals are reported as percentages (number of infants per 100); Difference in proportions = -3.0, 95% CI 2-sided [-5.4 to -0.4]
Statistical Analysis 8: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 7]; Difference in proportions = 1.4, 95% CI 2-sided [-0.6 to 4.8]

2. Primary Outcome: Number of Participants With Seroprotection for Meningitis Serogroup X (NmCV-5) vs Lowest Comparator (MenACWY-TT)
Description: Null hypothesis: At Day 29, the immune response to meningitis serogroup X elicited by one dose of NmCV-5 is inferior to the lowest immune response (among meningitis serogroups A, C, W or Y) elicited by one dose of MenACWY-TT.
  Alternative hypothesis: At Day 29, the immune response to meningitis serogroup X elicited by one dose of NmCV-5 is non-inferior, by a pre-specified margin, to the lowest immune response (among meningitis serogroups A, C, W or Y) elicited by one dose of MenACWY-TT.
  Endpoints are the seroprotective response to serogroup X in the NmCV-5 arm and the minimum seroprotective response among serogroups A, C, W and Y in the MenACWY-TT arm at Day 29 with seroprotective response defined as serogroup specific rSBA antibody titers ≥ 8.
  Non-inferiority comparisons are made between study vaccination arms within each study age group (9 months or 15 months).
  Proportions and difference in proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 372 | 191 | 367 | 182
Participants
  Participants with seroprotective response against serogroup X (NmCV-5) and serogroup W (MenACWY-TT): number analyzed (Participants) | 372 | 191 | 0 | 0
  Participants with seroprotective response against serogroup X (NmCV-5) and serogroup W (MenACWY-TT): Yes | 371 | 186 |  |
  Participants with seroprotective response against serogroup X (NmCV-5) and serogroup W (MenACWY-TT): No | 1 | 5 |  |
  Participants with seroprotective response against serogroup X (NmCV-5) and serogroup Y (MenACWY-TT): number analyzed (Participants) | 0 | 0 | 367 | 182
  Participants with seroprotective response against serogroup X (NmCV-5) and serogroup Y (MenACWY-TT): Yes |  |  | 366 | 178
  Participants with seroprotective response against serogroup X (NmCV-5) and serogroup Y (MenACWY-TT): No |  |  | 1 | 4
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For the 9-months study age group, the proportion of infants with a seroprotective response to MenACWY-TT in serogroup W is subtracted from the proportion of infants with a seroprotective response to NmCV-5 in serogroup X to determine the difference in proportions; Test type: Non-Inferiority — NmCV-5 will be deemed non-inferior to MenACWY-TT for serogroup X if the lower limit of the 95% confidence interval (CI) for the difference in proportion (NmCV-5 minus MenACWY-TT) excludes -0.10 (-10%). The CI is estimated using bootstrap resampling stratified by vaccine arm, and the 95% CI is estimated as the interval between the 2.5th and 97.5th percentiles of the bootstrap empirical distribution. The difference in proportions and CI are reported as percentages (number of infants per 100); Difference in proportions = 2.3, 95% CI 2-sided [0.3 to 4.7]
Statistical Analysis 2: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; For the 15-months study age group, the proportion of infants with a seroprotective response to MenACWY-TT in serogroup Y is subtracted from the proportion of infants with a seroprotective response to NmCV-5 in serogroup X to determine the difference in proportions; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in proportions = 1.9, 95% CI 2-sided [0.004 to 4.4]

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: To assess the safety and tolerability of a single dose of NmCV-5 or MenACWY-TT, when given concomitantly with routine vaccines, all Serious Adverse Events (SAE) occurring during the first 6 months of the follow-up period after meningococcal vaccination are reported.
  Endpoints are the number of participants with unsolicited adverse events that are reported as Serious Adverse Events (SAEs) according to ICH/GCP guidelines or the study protocol collected from the time of Step 2 randomization and vaccination and with date of event onset up to and including Study Day 181.
Time Frame: Measured from time of meningococcal vaccination to Study Day 181 or early study termination, whichever is earlier. Follow-up time to Study Day 181 visit was a mean (s.d.) of 180.8 (3.0) days.
Population: All participants included in the modified intent-to-treat (mITT) Analysis Set which includes all participants who were randomized at Step 1 and Step 2 and who received a study meningitis vaccine (NmCV-5 or MenACWY-TT).
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 400 | 200 | 400 | 200
Participants
  Participants experiencing SAE: Yes | 1 | 0 | 2 | 1
  Participants experiencing SAE: No | 399 | 200 | 398 | 199
  Gastroenteritis: Yes | 0 | 0 | 1 | 0
  Gastroenteritis: No | 400 | 200 | 399 | 200
  Thermal burn: Yes | 0 | 0 | 1 | 1
  Thermal burn: No | 400 | 200 | 399 | 199
  Malnutrition: Yes | 1 | 0 | 0 | 0
  Malnutrition: No | 399 | 200 | 400 | 200

4. Secondary Outcome: Number of Participants With Solicited Adverse Events (Reactogenicity)
Description: To assess the safety and tolerability of a single dose of NmCV-5 or MenACWY-TT, when given concomitantly with routine vaccines, all solicited AEs occurring during a 7-day follow-up period after meningococcal vaccination are reported. Solicited AEs include injection site (local) events (erythema/redness, induration/swelling, pain and/or tenderness) and systemic events (irritability, drowsiness/lethargy, decrease eating/anorexia, vomiting, fever (axillary), and feverish).
  Endpoints are the number of participants with solicited adverse events collected from about 30 minutes after meningococcal vaccination to Study Day 8 (7 days after vaccination).
  NOTE: Capture of data for symptom Feverish began on June 15, 2022, so some participants were not assessed for this symptom. Also, Fever (Axillary) is objectively measured by oral temperature and Feverish is a subjective observation from a parent who feels their infant has a raised temperature but not verified by thermometer.
Time Frame: Measured from about 30 minutes after meningococcal vaccination to Study Day 8 (7 days) for all participants.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 400 | 200 | 400 | 200
Participants
  Participants experiencing a solicited AE: Yes | 250 | 137 | 115 | 45
  Participants experiencing a solicited AE: No | 150 | 63 | 285 | 155
  Participants experiencing a solicited AE: Not Evaluated | 0 | 0 | 0 | 0
  Participants experiencing a local solicited AE: Yes | 238 | 129 | 106 | 44
  Participants experiencing a local solicited AE: No | 162 | 71 | 294 | 156
  Participants experiencing a local solicited AE: Not Evaluated | 0 | 0 | 0 | 0
  Erythema/redness: Yes | 1 | 3 | 0 | 0
  Erythema/redness: No | 399 | 197 | 400 | 200
  Erythema/redness: Not Evaluated | 0 | 0 | 0 | 0
  Induration/swelling: Yes | 48 | 31 | 2 | 0
  Induration/swelling: No | 352 | 169 | 398 | 200
  Induration/swelling: Not Evaluated | 0 | 0 | 0 | 0
  Pain and/or tenderness: Yes | 224 | 120 | 106 | 44
  Pain and/or tenderness: No | 176 | 80 | 294 | 156
  Pain and/or tenderness: Not Evaluated | 0 | 0 | 0 | 0
  Participants experiencing a systemic solicited AE: Yes | 60 | 32 | 16 | 3
  Participants experiencing a systemic solicited AE: No | 340 | 168 | 384 | 197
  Participants experiencing a systemic solicited AE: Not Evaluated | 0 | 0 | 0 | 0
  Irritability: Yes | 17 | 5 | 3 | 1
  Irritability: No | 383 | 195 | 397 | 199
  Irritability: Not Evaluated | 0 | 0 | 0 | 0
  Drowsiness/lethargy: Yes | 4 | 2 | 3 | 1
  Drowsiness/lethargy: No | 396 | 198 | 397 | 199
  Drowsiness/lethargy: Not Evaluated | 0 | 0 | 0 | 0
  Decrease eating/anorexia: Yes | 2 | 0 | 4 | 1
  Decrease eating/anorexia: No | 398 | 200 | 396 | 199
  Decrease eating/anorexia: Not Evaluated | 0 | 0 | 0 | 0
  Vomiting: Yes | 4 | 3 | 5 | 1
  Vomiting: No | 396 | 197 | 395 | 199
  Vomiting: Not Evaluated | 0 | 0 | 0 | 0
  Fever (axillary): Yes | 6 | 5 | 3 | 2
  Fever (axillary): No | 394 | 195 | 397 | 198
  Fever (axillary): Not Evaluated | 0 | 0 | 0 | 0
  Feverish: Yes | 41 | 20 | 7 | 2
  Feverish: No | 147 | 73 | 393 | 198
  Feverish: Not Evaluated | 212 | 107 | 0 | 0

5. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: To assess the safety and tolerability of a single dose of NmCV-5 or MenACWY-TT, when given concomitantly with routine vaccines, all unsolicited AEs occurring through 28 days after meningococcal vaccination are reported. Unsolicited AEs include AEs reported in scheduled or interim (unscheduled) visits after receipt of meningitis vaccination and with date of onset up to and including Study Day 29.
  Endpoints are the number of participants reporting at least one unsolicited adverse event (overall and by MedDRA preferred term).
Time Frame: Measured from time of meningococcal vaccination to Study Day 29 (28 days) for all participants.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 400 | 200 | 400 | 200
Participants
  Participants experiencing an unsolicited AE: Yes | 64 | 37 | 16 | 8
  Participants experiencing an unsolicited AE: No | 336 | 163 | 384 | 192
  Allergic cough: Yes | 1 | 0 | 0 | 0
  Allergic cough: No | 399 | 200 | 400 | 200
  Bronchitis: Yes | 10 | 13 | 4 | 3
  Bronchitis: No | 390 | 187 | 396 | 197
  Conjunctivitis: Yes | 0 | 0 | 1 | 1
  Conjunctivitis: No | 400 | 200 | 399 | 199
  Diarrhoea: Yes | 19 | 7 | 1 | 1
  Diarrhoea: No | 381 | 193 | 399 | 199
  Gastroenteritis: Yes | 5 | 3 | 4 | 0
  Gastroenteritis: No | 395 | 197 | 396 | 200
  Impetigo: Yes | 4 | 4 | 0 | 0
  Impetigo: No | 396 | 196 | 400 | 200
  Malaria: Yes | 1 | 0 | 0 | 0
  Malaria: No | 399 | 200 | 400 | 200
  Nasopharyngitis: Yes | 2 | 2 | 0 | 0
  Nasopharyngitis: No | 398 | 198 | 400 | 200
  Otitis media acute: Yes | 1 | 1 | 0 | 0
  Otitis media acute: No | 399 | 199 | 400 | 200
  Otorrhoea: Yes | 2 | 0 | 0 | 0
  Otorrhoea: No | 398 | 200 | 400 | 200
  Pharyngitis: Yes | 9 | 5 | 5 | 2
  Pharyngitis: No | 391 | 195 | 395 | 198
  Pyoderma: Yes | 9 | 3 | 0 | 0
  Pyoderma: No | 391 | 197 | 400 | 200
  Rhinitis: Yes | 5 | 2 | 2 | 1
  Rhinitis: No | 395 | 198 | 398 | 199

6. Secondary Outcome: Number of Participants With Seroprotection for Meningitis Serogroup X
Description: Null hypothesis: The immune response to meningitis serogroup X at Day 29 elicited by one dose of NmCV-5 is not superior to the immune response elicited by one dose of MenACWY-TT, Alternative hypothesis: The immune response to meningitis serogroup X at Day 29 elicited by one dose of NmCV-5 is superior, by a pre-specified margin, to the immune response elicited by one dose of MenACWY-TT.
  Endpoints are the seroprotective response to serogroup X in the NmCV-5 arm at Day 29 and the seroprotective response defined to serogroup X in the MenACWY-TT arm at Day 29 with seroprotective response defined as serogroup specific rSBA antibody titers ≥ 8.
  Superiority comparisons are made between study vaccination arms within each study age group (9 months or 15 months of age).
  Proportions and difference in proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 372 | 191 | 367 | 182
Participants
  Yes | 371 | 33 | 366 | 57
  No | 1 | 158 | 1 | 125
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup X, the proportion of infants with a seroprotective response to MenACWY-TT is subtracted from the proportion of infants with a seroprotective response to NmCV-5 to determine the difference in proportions; Test type: Superiority — NmCV-5 will be deemed superior to MenACWY-TT for serogroup X if the lower limit of the 95% confidence interval for the difference in proportion (NmCV-5 minus MenACWY-TT) excludes 0.30 (30%). Confidence Intervals are calculated using the Miettinen-Nurminen method. The difference in proportions and CI are reported as percentages (number of infants per 100); Difference in proportions = 82.5, 95% CI 2-sided [76.4 to 87.2]
Statistical Analysis 2: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 6, analysis 1]; Test type: Superiority — [test comment as in outcome 6, analysis 1]; Difference in proportions = 68.4, 95% CI 2-sided [61.3 to 74.7]

7. Secondary Outcome: Number of Participants With Seropositive Response to Measles Vaccine
Description: Null hypothesis: The immune response to measles at Day 29 elicited by the MR vaccine when co-administered with one dose of NmCV-5 is inferior to the immune response elicited by the MR vaccine when co-administered with one dose of MenACWY-TT.
  Alternative hypothesis: The immune response to measles at Day 29 elicited by the MR vaccine when co-administered with one dose of NmCV-5 is non inferior, by a pre-specified margin, to the immune response elicited by the MR vaccine when co-administered with one dose of MenACWY-TT.
  Endpoints are the seropositive responses to measles vaccine at Day 29 post vaccination, defined as anti-measles IgG concentration >200 mIU/mL.
  Non-inferiority comparisons are made between study vaccination arms within each study age group (9 months or 15 months of age).
  Proportions and difference in proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 364 | 187 | 364 | 176
Participants
  Yes | 364 | 187 | 364 | 176
  No | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For this comparison, the proportion of infants with a seropositive response to measles vaccine in the MenACWY-TT arm is subtracted from the proportion of infants with a seropositive response to measles vaccine in the NmCV-5 arm to determine the difference in proportions; Test type: Non-Inferiority — The NmCV-5 co-administered MR vaccine will be deemed non-inferior to the MenACWY-TT co-administered MR vaccine in eliciting seropositive response to measles if the lower limit of the 95% confidence interval for the difference in proportions excludes -0.10 (-10%). Confidence Intervals are calculated using the Miettinen-Nurminen method. The difference in proportions and CI are reported as percentages (number of infants per 100); Difference in proportions = 0.0, 95% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 2: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; Difference in proportions = 0.0, 95% CI 2-sided [-1.0 to 2.1]

8. Secondary Outcome: Number of Participants With Seropositive Response to Rubella Vaccine
Description: Null hypothesis: The immune response to rubella at Day 29 elicited by the MR vaccine when co-administered with one dose of NmCV-5 is inferior to the immune response elicited by the MR vaccine when co-administered with one dose of MenACWY-TT.
  Alternative hypothesis: The immune response to rubella at Day 29 elicited by the MR vaccine when co-administered with one dose of NmCV-5 is non inferior, by a pre-specified margin, to the immune response elicited by the MR vaccine when co-administered with one dose of MenACWY-TT.
  Endpoints are the seropositive responses to rubella vaccine at Day 29 post vaccination, defined as anti-rubella IgG concentration >20 IU/mL.
  Non-inferiority comparisons are made between study vaccination arms within each study age group (9 months or 15 months of age).
  Proportions and difference in proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 364 | 187 | 364 | 176
Participants
  Yes | 294 | 159 | 364 | 176
  No | 70 | 28 | 0 | 0
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For this comparison, the proportion of infants with a seropositive response to rubella vaccine in the MenACWY-TT arm is subtracted from the proportion of infants with a seropositive response to rubella vaccine in the NmCV-5 arm to determine the difference in proportions; Test type: Non-Inferiority — The NmCV-5 co-administered MR vaccine will be deemed non-inferior to the MenACWY-TT co-administered MR vaccine in eliciting seropositive response to rubella if the lower limit of the 95% confidence interval for the difference in proportions excludes -0.10 (-10%). Confidence Intervals are calculated using the Miettinen-Nurminen method. The difference in proportions and CI are reported as percentages (number of infants per 100); Difference in proportions = -4.3, 95% CI 2-sided [-10.5 to 2.6]
Statistical Analysis 2: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; Difference in proportions = 0.0, 95% CI 2-sided [-1.0 to 2.1]

9. Secondary Outcome: Number of Participants With Seroprotective Response to Yellow Fever Vaccine
Description: Null hypothesis: The immune response to yellow fever at Day 29 elicited by the yellow fever vaccine when co-administered with one dose of NmCV-5 is inferior to the immune response elicited by the yellow fever vaccine when co-administered with one dose of MenACWY-TT.
  Alternative hypothesis: The immune response to yellow fever at Day 29 elicited by the yellow fever vaccine when co-administered with one dose of NmCV-5 is non inferior, by a pre-specified margin, to the immune response elicited by the yellow fever vaccine when co-administered with one dose of MenACWY-TT.
  Endpoints are the seroprotective responses to yellow fever vaccine at Day 29 post vaccination, defined as yellow fever neutralizing antibody titers ≥10.
  Non-inferiority comparisons are made between study vaccination arms within the 9 months study age group only.
  Proportions and difference in proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 1
Population: All Group 1 participants included in the Per Protocol (PP) Analysis Set which includes eligible participants receiving step 1 and 2 randomizations, the randomized meningococcal vaccination in the appropriate age group window with the scheduled EPI vaccinations, and who had a blood specimen collected in the appropriate window around the Day 29 visit and a successful rSBA value provided by the laboratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 364 | 187 | 0 | 0
Participants
  Yes | 355 | 186 |  |
  No | 9 | 1 |  |
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For this comparison, the proportion of infants with a seroprotective response to yellow fever vaccine in the MenACWY-TT arm is subtracted from the proportion of infants with a seroprotective response to yellow fever vaccine in the NmCV-5 arm to determine the difference in proportions; Test type: Non-Inferiority — The NmCV-5 co-administered yellow fever vaccine will be deemed non-inferior to the MenACWY-TT co-administered yellow fever vaccine in eliciting seroprotective response to yellow fever if the lower limit of the 95% confidence interval for the difference in proportions excludes -0.10 (-10%). Confidence Intervals are calculated using the Miettinen-Nurminen method. The difference in proportions and CI are reported as percentages (number of infants per 100); Difference in proportions = -1.9, 95% CI 2-sided [-4.2 to 0.6]

10. Secondary Outcome: Geometric Mean of rSBA Titers for Meningitis Serogroups A, C, W, Y and X
Description: For each study age group (9 months and 15 months) and for each of the five serogroups (A, C, W, Y, and X), geometric means and 95% CIs of rSBA titers at Day 29 are calculated by study vaccination arm within each study age group, and the Geometric Mean Titer (GMT) Ratio of rSBA titers at Day 29 for NmCV-5 relative to MenACWY-TT will be estimated, along with 95% CIs. The point and interval estimates will be obtained from a back transformation of the estimated difference in means of the log-transformed rSBA titers.
  Endpoints are the rSBA titer values for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 3 (Study Day 29).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: rSBA titer
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 373 | 191 | 367 | 182
rSBA titer
  Serogroup A | 8131.3 [7187.9 to 9198.6] | 7814.5 [6706.2 to 9105.9] | 13436.7 [11822.1 to 15271.9] | 10942.0 [8774.4 to 13644.9]
  Serogroup C | 738.3 [636.1 to 857.0] | 1565.7 [1296.1 to 1891.4] | 807.1 [689.2 to 945.2] | 2103.3 [1705.4 to 2594.2]
  Serogroup W | 2612.5 [2034.2 to 3355.1] | 2933.3 [2281.1 to 3772.0] | 7383.7 [6159.8 to 8850.9] | 4733.8 [3634.4 to 6165.8]
  Serogroup Y | 2086.4 [1731.6 to 2514.0] | 2798.2 [2350.1 to 3331.7] | 3629.6 [3208.7 to 4105.9] | 3598.5 [2848.6 to 4545.8]
  Serogroup X: number analyzed (Participants) | 372 | 191 | 367 | 182
  Serogroup X | 7352.8 [6640.7 to 8141.4] | 4.9 [3.6 to 6.6] | 9262.0 [8244.3 to 10405.3] | 12.1 [8.1 to 18.1]
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup A, the point and interval estimates for the Geometric Mean Titer (GMT) ratio will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMT ratio of rSBA titers at Day 29 is calculated for the NmCV-5 arm relative to the MenACWY-TT arm; Test type: Other; Ratio of geometric mean titers = 1.0, 95% CI 2-sided [0.8 to 1.3] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 2: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 10, analysis 1]; Test type: Other; Ratio of geometric mean titers = 1.2, 95% CI 2-sided [1.0 to 1.6] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 3: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup C, the point and interval estimates for the Geometric Mean Titer (GMT) ratio will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMT ratio of rSBA titers at Day 29 is calculated for the NmCV-5 arm relative to the MenACWY-TT arm; Test type: Other; Ratio of geometric mean titers = 0.5, 95% CI 2-sided [0.4 to 0.6] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 4: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 10, analysis 3]; Test type: Other; Ratio of geometric mean titers = 0.4, 95% CI 2-sided [0.3 to 0.5] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 5: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup W, the point and interval estimates for the Geometric Mean Titer (GMT) ratio will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMT ratio of rSBA titers at Day 29 is calculated for the NmCV-5 arm relative to the MenACWY-TT arm; Test type: Other; Ratio of geometric mean titers = 0.9, 95% CI 2-sided [0.6 to 1.3] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 6: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 10, analysis 5]; Test type: Other; Ratio of geometric mean titers = 1.6, 95% CI 2-sided [1.1 to 2.1] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 7: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup Y, the point and interval estimates for the Geometric Mean Titer (GMT) ratio will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMT ratio of rSBA titers at Day 29 is calculated for the NmCV-5 arm relative to the MenACWY-TT arm; Test type: Other; Ratio of geometric mean titers = 0.7, 95% CI 2-sided [0.6 to 1.0] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 8: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 10, analysis 7]; Test type: Other; Ratio of geometric mean titers = 1.0, 95% CI 2-sided [0.8 to 1.3] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 9: Comparison: Vaccination at 9 Months of Age With NmCV-5 vs Vaccination at 9 Months of Age With MenACWY-TT; For serogroup X, the point and interval estimates for the Geometric Mean Titer (GMT) ratio will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMT ratio of rSBA titers at Day 29 is calculated for the NmCV-5 arm relative to the MenACWY-TT arm; Test type: Other; Ratio of geometric mean titers = 1511.1, 95% CI 2-sided [1169.5 to 1952.4] — NmCV-5 divided by MenACWY-TT
Statistical Analysis 10: Comparison: Vaccination at 15 Months of Age With NmCV-5 vs Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 10, analysis 9]; Test type: Other; Ratio of geometric mean titers = 767.3, 95% CI 2-sided [553.2 to 1064.4] — NmCV-5 divided by MenACWY-TT

11. Secondary Outcome: Seroresponse for Meningitis Serogroups A, C, W, Y and X
Description: To assess clinically significant immune response indicators elicited by a single dose of meningococcal vaccine, the number and proportion of participants with seroresponse in rSBA titers at Day 29 is calculated for meningococcal serogroups A, C, W, Y and X.
  Endpoints are the number and percentage of participants with seroresponse in rSBA titers to meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 3 (Study Day 29), where seroresponse is defined as a post-immunization (Day 29) rSBA titer of 32 or greater if the participant's pre-immunization (Baseline) rSBA titer was < 8; or a ≥ four-fold increase over baseline at Day 29 post-immunization if the participant's pre-immunization rSBA titer was ≥ 8.
  Seroresponse is calculated for each study vaccination arm within each study age group (9 months or 15 months of age).
  Proportions are reported as percentages (number of infants per 100).
Time Frame: Measured from time of blood sample collection just prior to meningococcal vaccination at Day 1 visit to blood sample collection at Day 29 visit. Follow-up time to Day 29 visit blood specimen collection was a mean (s.d.) of 30.9 (2.8) days.
Population: All participants included in the Baseline Immunogenicity Analysis Set which includes a subset of participants randomly selected for assessment of baseline rSBA titers from blood samples collected at Day 1 (pre-vaccination). This set includes up to 150 participants from Group 1 and 198 participants from Group 2 who had a blood specimen collected in the appropriate window around the Day 29 visit and a successful rSBA value provided by the laboratory for both the Day 1 and Day 29 visit samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 98 | 48 | 118 | 61
Participants
  Participants with Serogroup A Seroresponse: Yes | 98 | 47 | 116 | 57
  Participants with Serogroup A Seroresponse: No | 0 | 1 | 2 | 4
  Participants with Serogroup C Seroresponse: Yes | 96 | 47 | 112 | 58
  Participants with Serogroup C Seroresponse: No | 2 | 1 | 6 | 3
  Participants with Serogroup W Seroresponse: Yes | 92 | 48 | 117 | 59
  Participants with Serogroup W Seroresponse: No | 6 | 0 | 1 | 2
  Participants with Serogroup Y Seroresponse: Yes | 94 | 48 | 117 | 57
  Participants with Serogroup Y Seroresponse: No | 4 | 0 | 1 | 4
  Participants with Serogroup X Seroresponse: number analyzed (Participants) | 97 | 48 | 118 | 61
  Participants with Serogroup X Seroresponse: Yes | 97 | 7 | 115 | 9
  Participants with Serogroup X Seroresponse: No | 0 | 41 | 3 | 52

12. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Meningitis Serogroups A, C, W, Y and X
Description: To assess clinically significant immune response indicators elicited by a single dose of meningococcal vaccine, the Geometric Mean Fold Rise (GMFR) from baseline to Day 29 of rSBA titers to meningococcal serogroups A, C, W, Y and X is estimated, with 95% CI.
  Endpoints are the rSBA titer values for meningococcal serogroups A, C, W, Y and X from samples collected at Visit 1 (Day 1) and Visit 3 (Day 29).
  The point and interval estimates will be obtained from a back transformation of the estimated mean difference of the log-transformed rSBA titers.
Time Frame: as for outcome 11
Population: Participants in the Baseline Immunogenicity Analysis Set include a subset of participants randomly selected for assessment of baseline rSBA titers from blood samples collected at Day 1 (pre-vaccination). This set includes up to 150 participants from Group 1 and 198 participants from Group 2 who had a blood specimen collected in the appropriate window around the Day 29 visit and a successful rSBA value provided by the laboratory for both the Day 1 and Day 29 visit samples.
Measure: Geometric Mean (95% Confidence Interval); unit: rSBA titer
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 100 | 50 | 132 | 66
rSBA titer
  Serogroup A, Day 1 | 2.6 [2.1 to 3.2] | 3.3 [2.0 to 5.5] | 10.6 [6.8 to 16.5] | 8.2 [4.5 to 14.7]
  Serogroup A, Day 29: number analyzed (Participants) | 98 | 48 | 118 | 61
  Serogroup A, Day 29 | 7111.4 [5538.4 to 9131.2] | 8554.7 [6613.9 to 11064.9] | 13817.8 [11112.3 to 17182.0] | 7917.4 [4920.2 to 12740.4]
  Serogroup C, Day 1 | 2.2 [2.0 to 2.4] | 2.4 [1.9 to 3.1] | 2.2 [2.0 to 2.5] | 2.3 [1.9 to 2.7]
  Serogroup C, Day 29: number analyzed (Participants) | 98 | 48 | 118 | 61
  Serogroup C, Day 29 | 633.0 [474.3 to 844.9] | 1602.2 [1039.7 to 2469.0] | 647.6 [488.0 to 859.4] | 1934.9 [1202.6 to 3113.1]
  Serogroup W, Day 1 | 2.2 [1.9 to 2.5] | 2.5 [1.8 to 3.3] | 2.4 [2.1 to 2.8] | 2.3 [1.9 to 2.8]
  Serogroup W, Day 29: number analyzed (Participants) | 98 | 48 | 118 | 61
  Serogroup W, Day 29 | 2326.1 [1504.8 to 3595.5] | 4801.2 [3587.7 to 6425.0] | 7770.2 [5686.2 to 10617.9] | 3226.5 [1934.9 to 5380.1]
  Serogroup Y, Day 1 | 2.4 [2.0 to 2.8] | 2.4 [1.9 to 3.0] | 5.7 [4.0 to 8.2] | 5.4 [3.1 to 9.2]
  Serogroup Y, Day 29: number analyzed (Participants) | 98 | 48 | 118 | 61
  Serogroup Y, Day 29 | 1908.2 [1326.1 to 2745.6] | 3494.4 [2505.3 to 4874.1] | 3454.4 [2783.3 to 4287.4] | 3083.1 [1848.0 to 5143.6]
  Serogroup X, Day 1 | 2.5 [2.1 to 3.1] | 2.2 [1.9 to 2.6] | 6.2 [4.2 to 9.1] | 8.3 [4.5 to 15.1]
  Serogroup X, Day 29: number analyzed (Participants) | 98 | 48 | 118 | 61
  Serogroup X, Day 29 | 6706.5 [5625.7 to 7995.0] | 4.4 [2.5 to 7.7] | 8687.6 [7142.1 to 10567.6] | 16.2 [7.6 to 34.4]
Statistical Analysis 1: Comparison: Vaccination at 9 Months of Age With NmCV-5; For serogroup A, the point and interval estimates for the Geometric Mean Fold Rise (GMFR) will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMFR from baseline to Day 29 of rSBA titers is calculated as Day 29 divided by Day 1; Test type: Other; Ratio of geometric mean titers = 2756.4, 95% CI 2-sided [1976.3 to 3844.5] — Day 29 divided by Day 1
Statistical Analysis 2: Comparison: Vaccination at 9 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 1]; Test type: Other; Ratio of geometric mean titers = 2506.9, 95% CI 2-sided [1404.0 to 4476.1] — Day 29 divided by Day 1
Statistical Analysis 3: Comparison: Vaccination at 15 Months of Age With NmCV-5; [analysis description as in outcome 12, analysis 1]; Test type: Other; Ratio of geometric mean titers = 1179.0, 95% CI 2-sided [709.8 to 1958.6] — Day 29 divided by Day 1
Statistical Analysis 4: Comparison: Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 1]; Test type: Other; Ratio of geometric mean titers = 1096.2, 95% CI 2-sided [513.4 to 2340.6] — Day 29 divided by Day 1
Statistical Analysis 5: Comparison: Vaccination at 9 Months of Age With NmCV-5; For serogroup C, the point and interval estimates for the Geometric Mean Fold Rise (GMFR) will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMFR from baseline to Day 29 of rSBA titers is calculated as Day 29 divided by Day 1; Test type: Other; Ratio of geometric mean titers = 288.7, 95% CI 2-sided [212.6 to 392.0] — Day 29 divided by Day 1
Statistical Analysis 6: Comparison: Vaccination at 9 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 5]; Test type: Other; Ratio of geometric mean titers = 654.5, 95% CI 2-sided [385.5 to 1111.0] — Day 29 divided by Day 1
Statistical Analysis 7: Comparison: Vaccination at 15 Months of Age With NmCV-5; [analysis description as in outcome 12, analysis 5]; Test type: Other; Ratio of geometric mean titers = 287.9, 95% CI 2-sided [213.9 to 387.5] — Day 29 divided by Day 1
Statistical Analysis 8: Comparison: Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 5]; Test type: Other; Ratio of geometric mean titers = 834.6, 95% CI 2-sided [496.7 to 1402.3] — Day 29 divided by Day 1
Statistical Analysis 9: Comparison: Vaccination at 9 Months of Age With NmCV-5; For serogroup W, the point and interval estimates for the Geometric Mean Fold Rise (GMFR) will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMFR from baseline to Day 29 of rSBA titers is calculated as Day 29 divided by Day 1; Test type: Other; Ratio of geometric mean titers = 1068.4, 95% CI 2-sided [683.3 to 1670.6] — Day 29 divided by Day 1
Statistical Analysis 10: Comparison: Vaccination at 9 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 9]; Test type: Other; Ratio of geometric mean titers = 1933.1, 95% CI 2-sided [1224.7 to 3051.1] — Day 29 divided by Day 1
Statistical Analysis 11: Comparison: Vaccination at 15 Months of Age With NmCV-5; [analysis description as in outcome 12, analysis 9]; Test type: Other; Ratio of geometric mean titers = 3163.1, 95% CI 2-sided [2247.5 to 4451.7] — Day 29 divided by Day 1
Statistical Analysis 12: Comparison: Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 9]; Test type: Other; Ratio of geometric mean titers = 1524.1, 95% CI 2-sided [913.5 to 2543.0] — Day 29 divided by Day 1
Statistical Analysis 13: Comparison: Vaccination at 9 Months of Age With NmCV-5; For serogroup Y, the point and interval estimates for the Geometric Mean Fold Rise (GMFR) will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMFR from baseline to Day 29 of rSBA titers is calculated as Day 29 divided by Day 1; Test type: Other; Ratio of geometric mean titers = 799.4, 95% CI 2-sided [532.9 to 1199.4] — Day 29 divided by Day 1
Statistical Analysis 14: Comparison: Vaccination at 9 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 13]; Test type: Other; Ratio of geometric mean titers = 1469.2, 95% CI 2-sided [995.3 to 2168.8] — Day 29 divided by Day 1
Statistical Analysis 15: Comparison: Vaccination at 15 Months of Age With NmCV-5; [analysis description as in outcome 12, analysis 13]; Test type: Other; Ratio of geometric mean titers = 549.4, 95% CI 2-sided [371.8 to 811.8] — Day 29 divided by Day 1
Statistical Analysis 16: Comparison: Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 13]; Test type: Other; Ratio of geometric mean titers = 642.6, 95% CI 2-sided [309.2 to 1335.9] — Day 29 divided by Day 1
Statistical Analysis 17: Comparison: Vaccination at 9 Months of Age With NmCV-5; For serogroup X, the point and interval estimates for the Geometric Mean Fold Rise (GMFR) will be obtained from a back transformation (exponentiation) of the estimated mean ratio of the log-transformed rSBA titers. The GMFR from baseline to Day 29 of rSBA titers is calculated as Day 29 divided by Day 1; Test type: Other; Ratio of geometric mean titers = 2630.0, 95% CI 2-sided [2037.6 to 3394.6] — Day 29 divided by Day 1
Statistical Analysis 18: Comparison: Vaccination at 9 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 17]; Test type: Other; Ratio of geometric mean titers = 2.0, 95% CI 2-sided [1.2 to 3.4] — Day 29 divided by Day 1
Statistical Analysis 19: Comparison: Vaccination at 15 Months of Age With NmCV-5; [analysis description as in outcome 12, analysis 17]; Test type: Other; Ratio of geometric mean titers = 1431.2, 95% CI 2-sided [905.2 to 2262.9] — Day 29 divided by Day 1
Statistical Analysis 20: Comparison: Vaccination at 15 Months of Age With MenACWY-TT; [analysis description as in outcome 12, analysis 17]; Test type: Other; Ratio of geometric mean titers = 1.7, 95% CI 2-sided [0.9 to 3.3] — Day 29 divided by Day 1

13. Secondary Outcome: Number of Participants With rSBA Titers ≥ 128 for Meningitis Serogroups A, C, W, Y and X
Description: To assess clinically significant immune response indicators elicited by a single dose of meningococcal vaccine, the number and proportion of participants with rSBA titers ≥ 128 at Day 29 is calculated for meningococcal serogroups A, C, W, Y and X.
  Endpoints are the number and proportion of participants with rSBA titers ≥ 128 for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 3 (Study Day 29).
  This is calculated for each study vaccination arm within each study age group (9 months or 15 months of age).
  Proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
Number analyzed (Participants) | 373 | 191 | 367 | 182
Participants
  Serogroup A, Participants with rSBA titer ≥ 128: Yes | 372 | 191 | 366 | 180
  Serogroup A, Participants with rSBA titer ≥ 128: No | 1 | 0 | 1 | 2
  Serogroup C, Participants with rSBA titer ≥ 128: Yes | 354 | 187 | 351 | 179
  Serogroup C, Participants with rSBA titer ≥ 128: No | 19 | 4 | 16 | 3
  Serogroup W, Participants with rSBA titer ≥ 128: Yes | 348 | 185 | 362 | 177
  Serogroup W, Participants with rSBA titer ≥ 128: No | 25 | 6 | 5 | 5
  Serogroup Y, Participants with rSBA titer ≥ 128: Yes | 356 | 190 | 364 | 178
  Serogroup Y, Participants with rSBA titer ≥ 128: No | 17 | 1 | 3 | 4
  Serogroup X, Participants with rSBA titer ≥ 128: number analyzed (Participants) | 372 | 191 | 367 | 182
  Serogroup X, Participants with rSBA titer ≥ 128: Yes | 371 | 29 | 366 | 51
  Serogroup X, Participants with rSBA titer ≥ 128: No | 1 | 162 | 1 | 131

14. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAE) Through 2 Years of Follow-Up
Description: To assess the safety and tolerability of a single dose of NmCV-5 or MenACWY-TT, when given concomitantly with routine vaccines, all Serious Adverse Events (SAE) occurring during 2 years of follow-up after meningococcal vaccination are reported.
  Endpoints are the number of participants with unsolicited adverse events that are reported as Serious Adverse Events (SAEs) according to ICH/GCP guidelines or the study protocol collected from the time of Step 2 randomization and vaccination and with date of event onset up to and including Study Day 730.
Time Frame: Measured from time of meningococcal vaccination to Study Day 730 or early study termination, whichever is earlier. Follow-up time to Study Day 730 visit was a mean (s.d.) of xxx.x (x.x) days.
Reporting Status: Not Posted, anticipated posting 2025-09

15. Other Pre Specified Outcome: Geometric Mean of rSBA Titers at Study Day 181 for Meningitis Serogroups A, C, W, Y and X
Description: For each study age group (9 months and 15 months) and for each of the five serogroups (A, C, W, Y, and X), geometric means and 95% CIs of rSBA titers at Day 181 are calculated by study vaccination arm within each study age group.
  Endpoints are the rSBA titer values for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 4 (Study Day 181).
Time Frame: Measured from time of meningococcal vaccination to blood sample collection at Day 181 visit. Follow-up time to Day 181 visit blood specimen collection was a mean (s.d.) of xx.x (x.x) days.
Reporting Status: Not Posted, anticipated posting 2025-09

16. Other Pre Specified Outcome: Number of Participants With rSBA Titers ≥ 8 at Study Day 181 for Meningitis Serogroups A, C, W, Y and X
Description: To assess the persistence of immune response elicited by a single dose of meningococcal vaccine, the number and proportion of participants with rSBA titers ≥ 8 at Day 181 is calculated for meningococcal serogroups A, C, W, Y and X.
  Endpoints are the number and proportion of participants with rSBA titers ≥ 8 for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 4 (Study Day 181).
  This is calculated for each study vaccination arm within each study age group (9 months or 15 months of age).
  Proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 15
Reporting Status: Not Posted, anticipated posting 2025-09

17. Other Pre Specified Outcome: Number of Participants With rSBA Titers ≥ 128 at Study Day 181 for Meningitis Serogroups A, C, W, Y and X
Description: To assess the persistence of immune response elicited by a single dose of meningococcal vaccine, the number and proportion of participants with rSBA titers ≥ 128 at Day 181 is calculated for meningococcal serogroups A, C, W, Y and X.
  Endpoints are the number and proportion of participants with rSBA titers ≥ 128 for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 4 (Study Day 181).
  This is calculated for each study vaccination arm within each study age group (9 months or 15 months of age).
  Proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 15
Reporting Status: Not Posted, anticipated posting 2025-09

18. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) at Study Day 181 for Meningitis Serogroups A, C, W, Y and X
Description: To assess the persistence of immune response elicited by a single dose of meningococcal vaccine, the Geometric Mean Fold Rise (GMFR) from baseline to Day 181 of rSBA titers to meningococcal serogroups A, C, W, Y and X is estimated, with 95% CI.
  Endpoints are the rSBA titer values for meningococcal serogroups A, C, W, Y and X from samples collected at Visit 1 (Day 1) and Visit 4 (Day 181).
  The point and interval estimates will be obtained from a back transformation of the estimated mean difference of the log-transformed rSBA titers.
Time Frame: Measured from time of blood sample collection just prior to meningococcal vaccination at Day 1 visit to blood sample collection at Day 181 visit. Follow-up time to Day 181 visit blood specimen collection was a mean (s.d.) of xx.x (x.x) days.
Reporting Status: Not Posted, anticipated posting 2025-09

19. Other Pre Specified Outcome: Geometric Mean of rSBA Titers at Study Day 730 for Meningitis Serogroups A, C, W, Y and X
Description: For each study age group (9 months and 15 months) and for each of the five serogroups (A, C, W, Y, and X), geometric means and 95% CIs of rSBA titers at Day 730 are calculated by study vaccination arm within each study age group.
  Endpoints are the rSBA titer values for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 5 (Study Day 730).
Time Frame: Measured from time of meningococcal vaccination to blood sample collection at Day 730 visit. Follow-up time to Day 730 visit blood specimen collection was a mean (s.d.) of xx.x (x.x) days.
Reporting Status: Not Posted, anticipated posting 2025-12

20. Other Pre Specified Outcome: Number of Participants With rSBA Titers ≥ 8 at Study Day 730 for Meningitis Serogroups A, C, W, Y and X
Description: To assess the persistence of immune response elicited by a single dose of meningococcal vaccine, the number and proportion of participants with rSBA titers ≥ 8 at Day 730 is calculated for meningococcal serogroups A, C, W, Y and X.
  Endpoints are the number and proportion of participants with rSBA titers ≥ 8 for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 5 (Study Day 730).
  This is calculated for each study vaccination arm within each study age group (9 months or 15 months of age).
  Proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 19
Reporting Status: Not Posted, anticipated posting 2025-12

21. Other Pre Specified Outcome: Number of Participants With rSBA Titers ≥ 128 at Study Day 730 for Meningitis Serogroups A, C, W, Y and X
Description: To assess the persistence of immune response elicited by a single dose of meningococcal vaccine, the number and proportion of participants with rSBA titers ≥ 128 at Day 730 is calculated for meningococcal serogroups A, C, W, Y and X.
  Endpoints are the number and proportion of participants with rSBA titers ≥ 128 for meningococcal serogroups A, C, W, Y and X, from samples collected at Visit 5 (Study Day 730).
  This is calculated for each study vaccination arm within each study age group (9 months or 15 months of age).
  Proportions are reported as percentages (number of infants per 100).
Time Frame: as for outcome 19
Reporting Status: Not Posted, anticipated posting 2025-12

22. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) at Study Day 730 for Meningitis Serogroups A, C, W, Y and X
Description: To assess the persistence of immune response elicited by a single dose of meningococcal vaccine, the Geometric Mean Fold Rise (GMFR) from baseline to Day 730 of rSBA titers to meningococcal serogroups A, C, W, Y and X is estimated, with 95% CI.
  Endpoints are the rSBA titer values for meningococcal serogroups A, C, W, Y and X from samples collected at Visit 1 (Day 1) and Visit 5 (Day 730).
  The point and interval estimates will be obtained from a back transformation of the estimated mean difference of the log-transformed rSBA titers.
Time Frame: Measured from time of blood sample collection just prior to meningococcal vaccination at Day 1 visit to blood sample collection at Day 730 visit. Follow-up time to Day 730 visit blood specimen collection was a mean (s.d.) of xx.x (x.x) days.
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) are recorded from the time of enrollment to Study Day 181. SAE follow-up time was approximately 6 months for participants receiving meningococcal vaccination at 9 months of age and for participants in Group 2 but not receiving meningococcal vaccination. SAE follow-up time was approximately 12 months for participants receiving vaccination at 15 months of age. Other non-serious AEs are reported from study vaccination through 28 days after vaccination(mITT population).
Description: SAEs were assessed for all 1325 participants who were enrolled and received step 1 randomization to Group 1 (9 months of age, n=602) or Group 2 (15 months of age, n=723, with n=600 further randomized and receiving meningococcal vaccine and n=123 not randomized and discontinued from the study). These 123 participants were followed for SAEs only during the pre-dosing period prior to step 2 randomization. Participants were routinely assessed for AEs at follow-up visits (Day 29, Day 181).
Arm/Group | Vaccination at 9 Months of Age With NmCV-5 | Vaccination at 9 Months of Age With MenACWY-TT | Not Vaccinated But Randomized to Vaccination at 15 Months of Age | Vaccination at 15 Months of Age With NmCV-5 | Vaccination at 15 Months of Age With MenACWY-TT
All-Cause Mortality (participants affected / at risk) | 0/401 | 0/201 | 1/123 | 0/400 | 0/200
Serious Adverse Events (participants affected / at risk) | 1/401 | 0/201 | 1/123 | 2/400 | 1/200
Other Adverse Events (participants affected / at risk) | 64/400 | 37/200 | 0/0 | 16/400 | 8/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccination at 9 Months of Age With NmCV-5 (N=401) | Vaccination at 9 Months of Age With MenACWY-TT (N=201) | Not Vaccinated But Randomized to Vaccination at 15 Months of Age (N=123) | Vaccination at 15 Months of Age With NmCV-5 (N=400) | Vaccination at 15 Months of Age With MenACWY-TT (N=200)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccination at 9 Months of Age With NmCV-5 (N=400) | Vaccination at 9 Months of Age With MenACWY-TT (N=200) | Not Vaccinated But Randomized to Vaccination at 15 Months of Age (N=0) | Vaccination at 15 Months of Age With NmCV-5 (N=400) | Vaccination at 15 Months of Age With MenACWY-TT (N=200)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 10 (10) | 13 (13) | NA | 4 (4) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | NA | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 19 (19) | 7 (7) | NA | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 3 (3) | NA | 4 (4) | 0 (0)
Impetigo (Infections and infestations) | 4 (4) | 4 (4) | NA | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | NA | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) | NA | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 2 (2) | 0 (0) | NA | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 9 (9) | 5 (5) | NA | 5 (5) | 2 (2)
Pyoderma (Infections and infestations) | 9 (9) | 3 (3) | NA | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 5 (5) | 2 (2) | NA | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT05093829/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT05093829/SAP_002.pdf
  • Informed Consent Form (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT05093829/ICF_000.pdf